CLINICAL TRIAL: NCT05053009
Title: The Effect of Ibuprofen Sustained Release Oral Premedication on Intraoperative and Postoperative Pain After Single-visit Root Canal Treatment of Mandibular Molars With Symptomatic Irreversible Pulpitis and Apical Periodontitis
Brief Title: Effect of Ibuprofen Sustained Release on Intraoperative and Postoperative Pain in Mandibular Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Ahmed Hossam, Resident at faculty of dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO3-7-1
Record Dates: First submitted 2021-09-11; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen sustained release (Experimental): Single dose of 800 mg Brufen Retard oral premedication will be administered 1 hour before local anesthesia
  Interventions: Drug: Brufen Retard
- Placebo (Placebo Comparator): 1 capsule of 500 mg of glucose oral premedication will be adminstered 1 hour before local anesthesia
  Interventions: Drug: Brufen Retard

INTERVENTIONS:
Drug: Brufen Retard — 800 mg tablet of Brufen Retard will be adminstered orally one hour before local anesthesia

SUMMARY:
The study is conducted to evaluate the effect of Ibuprofen sustained release premedication on the success of buccal infiltration anaesthesia, intaroperative pain and post operative pain in mandibular molars with symptomatic irreversible pulpitis and apical periodontitis

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy patients (ASA I or II).
2. Patients with Mandibular molar teeth diagnosed with:

   * Pre-operative sharp pain marked on VAS scale by reading not less than 6.
   * Vital exaggerated response of pulp tissue to cold pulp tester (ethyl chloride spray) and electric pulp tester.
   * Normal periapical radiographic appearance or slight widening in lamina dura.
   * Positive response and pain provoked by percussion.

Exclusion Criteria:

1. Allergy to Ibuprofen
2. Medically compromised patients having significant systemic disorders. (ASA III or IV).
3. History of intolerance to NSAIDS.
4. Patients with two or more adjacent teeth requiring endodontic treatment.
5. Pregnant or nursing females.
6. Teeth that have:

   * Periodontal affection (with pocket depth greater than 5mm, associated with swelling or fistulous tract, or greater than grade I mobility)
   * No possible restorability.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of buccal infiltration anaesthesia measured using Visual analogue scale | During root canal treatment procedures
  intensity of pain during root canal treatment procedures is recorded by the patient using VAS where 0=no pain, 1-3=mild pain, 4-6=moderate pain and 7-10=severe pain

SECONDARY OUTCOMES:
Intensity of intraoperative pain | During root canal treatment procedures
  intensity of pain during root canal treatment procedures is recorded by the patient using VAS where 0=no pain, 1-3=mild pain, 4-6=moderate pain and 7-10=severe pain
Postoperative pain | up to 48 hours after endodontic treatment
  Intensity of pain felt after endodontic treatment recorded by the patient using VAS where 0=no pain, 1-3=mild pain, 4-6=moderate pain and 7-10=severe pain
Number of needed analgesic tablets in case of intolerable pain | up to 48 hours after endodontic treatment
  The patient will record the number of analgesic tablets taken in case of intolerable pain